CLINICAL TRIAL: NCT06355713
Title: Prospective Multicenter Study of the Improvement of Symptoms After Removal of the Essure® Contraceptive Implant
Brief Title: Improvement of Symptoms After Removal of the Essure® Contraceptive Implant
Acronym: ABLES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0899; 2023-A02010-45 (Other: ID-RCB)
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Implant Complication; Contraceptive Device; Complications
Keywords: Essure implant; Contraceptive implant; Symptoms
MeSH Terms: interventions — Physical Examination; Blood Specimen Collection; Urine Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essure Group (Experimental): Patients requiring removal of the Essure® contraceptive implant
  Interventions: Device: Magnetic resonance imaging- Positron Emission Tomography (MRI-PET) examination; Biological: blood sample; Biological: urine collection; Biological: Collection of a lock of hair; Other: questionnaire
- Control Group (Active Comparator): Control patients who should benefit from a salpingectomy with or without hysterectomy for a benign indication
  Interventions: Device: Magnetic resonance imaging- Positron Emission Tomography (MRI-PET) examination; Biological: blood sample; Biological: urine collection; Biological: Collection of a lock of hair; Other: questionnaire

INTERVENTIONS:
Device: Magnetic resonance imaging- Positron Emission Tomography (MRI-PET) examination — An MRI-PET examination will be carried out pre-operatively and at 6 months for the first 20 patients with Essure® and pre-operatively for the first 10 control patients presenting the selection criteria.
  The duration of each acquisition will be approximately 2 hours. Upon arrival, participants will be greeted by electroradiography technicians. A venous catheter will be placed in a vein in the right or left arm. Participants will be installed in the hybrid MRI-PET imager. The injection of [11C]PK11195 will take place in the MRI-PET acquisition room. Recording of functional neuroimaging data will begin immediately after intravenous injection of [11C]PK11195 and will last for 70 minutes in a resting state.
  At the end of the examination, the venous catheter will be removed and the visit will be over.
Biological: blood sample — Patients with Essure : Blood sample pre-operatively (20 mL) and at 2 months (10 mL) and 12 months (5 mL).
  Control patients : Blood sample pre-operatively (20 mL)
Biological: urine collection — Patients with Essure : urine collection pre-operatively (10 mL) and at 2 months (10 mL) and 12 months (10 mL).
  Control patients : urine collection pre-operatively (10 mL)
Biological: Collection of a lock of hair — Patients with Essure : Collection of a lock of hair pre-operatively and at 12 months Control patients : Collection of a lock of hair pre-operatively
Other: questionnaire — Questionnaires pre-operatively (except PGI-I) and at 2, 6, 12 months then twice a year up to 5 years for patients with Essure, and pre-operatively (except PGI-I) and at 2 months for control patients :
  * PGI-I: symptom improvement score
  * SF-12: quality of life with physical and mental dimension.
  * FIQ: quality of life of women with fibromyalgia symptoms
  * HADS: anxiety and depressive dimension
  * MFI-20: fatigue according to 5 dimensions )
  * VAS : pain assessment
  * QDSA: assessment of sensory and emotional impact of pain
  * FSFI : quality of sexual life
  * Higham score

SUMMARY:
ESSURE® is an implantable medical device for definitive and irreversible sterilization indicated for adult women of childbearing age. These implants are inserted into the fallopian tubes by hysteroscopy. Marketed in 2002, ESSURE® contraceptive implants were withdrawn from the French market in 2017 (and worldwide in 2017 and 2018) following the observation in certain patients of polymorphic and non-specific gynecological and extra-gynecological symptoms. Studies with small numbers and short-term follow-up have shown a significant improvement in these symptoms after implant explantation. This constitutes a real public health problem since according to the report of the EPI-PHARE Scientific Interest Group, 198,000 French women have these implants and only 30,000 of them, or 15%, have been explanted, knowing that explantation of ESSURE® implants is recommended only in symptomatic patients. A large number of these patients, presenting symptoms, have not yet been treated for an explant.

The physiopathological mechanism(s) is (are) not yet determined but several arguments are in favor of a dissemination of metallic elements contained in these implants whose accumulation could lead to inflammatory and/or allergic and/or autoimmune phenomena.

Carrying out a prospective study with long-term longitudinal follow-up appears essential to precisely assess the degree of improvement in the symptoms and quality of life of these patients, determine the most appropriate surgical techniques, and understand the pathophysiological mechanisms that may result in the implementation of specific treatments and relevant markers. From a surgical point of view, there is a real risk of fracture of implants whatever the type of intervention performed: study the biomechanical properties of implants with a view to characterizing their behavior to mechanical rupture but also their thermal resistance in an objective manner seems essential to limit the risk of fracture and help to inform the patient about the surgical technique proposed for explantation. From a biological point of view, the dosage of the metallic elements constituting ESSURE® implants and potentially toxic ones could make it possible to objectify the release of these metallic elements in the body. Analysis of pro-inflammatory cytokines, micro-RNAs (miRNA), quantitative analysis of inflammatory pathway messenger ribonucleic acid (mRNAs) (NanoString technology) and analysis of neuroinflammation by functional imaging should make it possible to explore potential pathophysiological mechanisms. This study responds to a significant request from patient associations.

ELIGIBILITY:
* Inclusion Criteria * :

ESSURE Group:

* woman aged 35 to 75
* patient with at least one Essure® implant
* surgical intervention planned because the patient is symptomatic: removal of the Essure® implant(s)
* planned intervention via vaginal route, laparoscopy, robotic surgery, or Transvaginal natural orifice transluminal endoscopic surgery (VNotes)
* patient having given free, informed and signed consent

Selection for MRI-PET examination:

* if the answer is "poor" or "bad" to the first question of the SF-12 pre-operatively
* no hysterectomy
* no analgesic treatment, or treatment stopped 48 hours before the examination
* no psychotropic treatment (anxiolytics, hypnotics (sleeping pills), antidepressants, mood stabilizers, neuroleptics)
* patient having given free, informed and signed consent

Control group:

* woman aged 35 to 75
* planned surgical intervention: salpingectomy with or without hysterectomy for benign indication
* planned intervention via vaginal route, laparoscopy, robotic surgery, or VNotes
* patient having given free, informed and signed consent

Selection for MRI-PET examination:

* age matching (+/- 5 years) with Essure® patients who have had an MRI-PET
* matching on surgical technique with Essure® patients who have had an MRI-PET: salpingectomy with or without hysterectomy
* no analgesic treatment, or treatment stopped 48 hours before the examination
* no psychotropic treatment (anxiolytics, hypnotics (sleeping pills), antidepressants, mood stabilizers, neuroleptics)
* patient having given free, informed and signed consent

  * Exclusion Criteria * :

ESSURE Group:

* asymptomatic patient
* planned intervention by laparotomy
* patient potentially exposed to other heavy metals: wearer of metallic orthopedic equipment (hip or knee prosthesis, etc.), wearer of coronary stent, or tubal ligation clip
* inability to understand the information given
* persons deprived of liberty by a judicial or administrative decision
* people undergoing psychiatric care
* people admitted to a health or social establishment for purposes other than research
* adults subject to a legal protection measure (guardianship, curatorship)
* people not affiliated to a social security scheme or beneficiaries of a similar scheme
* person participating in another interventional research that may interfere with the research

Selection for MRI-PET examination:

* claustrophobia
* dosimetry of all radiological examinations over the past year not acceptable

Control Group :

* current pregnancy
* patient with cancer
* patient who has already had an Essure® implant removed
* patient potentially exposed to heavy metals: wearer of metallic orthopedic equipment (hip or knee prosthesis, etc.), wearer of coronary stent, or tubal ligation clip
* planned intervention by laparotomy
* inability to understand the information given
* persons deprived of liberty by a judicial or administrative decision
* people undergoing psychiatric care
* people admitted to a health or social establishment for purposes other than research
* adults subject to a legal protection measure (guardianship, curatorship)
* people not affiliated to a social security scheme or beneficiaries of a similar scheme
* person participating in another interventional research that may interfere with the research

Selection for MRI-PET examination:

* claustrophobia
* dosimetry of all radiological examinations over the past year not acceptable

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 444 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2032-04-17 (Estimated); Study Completion 2037-02-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with improvement in symptoms Percentage of patients with improvement in symptoms | At 2 months after surgical intervention (removal of the Essure® contraceptive implant)
  Percentage of patients with a score of 1, 2 or 3 (corresponding to improvement in symptoms) on the Patient Global Impression of Improvement (PGI-I) scale.
  The PGI-I is a transition scale that is a single question asking the patient to rate their symptoms now, as compared with how it was prior to before beginning treatment on a scale from 1 = Very much better to 7 = Very much worse.

SECONDARY OUTCOMES:
Percentage of patients with improvement in symptoms | up 5 years
  Percentage of patients with a score of 1, 2 or 3 (corresponding to improvement in symptoms) on the PGI-I scale.
  The PGI-I is a transition scale that is a single question asking the patient to rate their symptoms now, as compared with how it was prior to before beginning treatment on a scale from 1 = Very much better to 7 = Very much worse.
Short Form 12 (SF-12) score | up 5 years
  quality of life with assessment of the physical dimension (from 9.94738 to 70.02246) and the mental dimension (from 5.89058 to 71.96825). For each, the average in the general population is 50.
Fibromyalgia Impact Questionnaire (FIQ) score | up 5 years
  quality of life of women with fibromyalgia symptoms (from 0 : no symptoms to 100 : important symptoms)
Hospital Anxiety and Depression scale (HADS) score | up 5 years
  anxiety dimension and depressive dimension (for each dimension, from 0 : no symptom to 21 : certain symptomatology)
Multidimensional Fatigue Inventory (MFI)-20 score | up 5 years
  Fatigue assessment according to 5 dimensions (General Fatigue, Physical and Mental Fatigue, Reduction in Motivation and Activities) (score from 20 : no fatigue to 100 : important fatigue)
Visual analog scale (VAS) score | up 5 years
  pain assessment (from 0 : no pain to 100 : unbearable pain)
Questionnaire Douleur St-Antoine (QDSA) score | up 5 years
  Assessment of sensory impact of pain (from 0: no pain to 36: important impact) and emotional impact of pain (from 0: no pain to 28 : important impact). The global score ranges from 0 to 64.
Female Sexual Function Index (FSFI) score | up 5 years
  quality of sexual life (from 2 to 36). A low score indicates poorer sexual function.
Higham questionnaires | up 5 years
  The Higham score is used to quantify blood loss during menstruation. A score ≥ 100 indicates a loss of 80 ml or more, which defines menorrhagia. A score ≥ 150 may indicate an indication for surgery for menometrorrhagia.
visual analog scale (VAS) score | During surgical intervention
  Assessment by the surgeon of the difficulty of performing the ablation on a visual analog scale : from 0 (very easy) to 100 mm (very difficult)
Duration of the procedure | During surgical intervention
  Duration of the procedure (calculated between incision and closure) in number of minutes
Complications | Up to 2 months after the operation
  Number and types of per- and post-operative complications
characterization of the mechanical behavior of the implant | During surgical intervention
  characterization of the mechanical behavior of the Essure® device implant will be assessed during tensile breakage and thermal breakage for its two parts (internal part and external part)
determination of the associated mechanical stress levels determination of the associated mechanical stress levels | During surgical intervention
  determination of the associated mechanical stress levels of the Essure® device implant will be assessed during tensile breakage and thermal breakage for its two parts (internal part and external part)
quantification of the factors influencing these levels of mechanical stress | During surgical intervention
  quantification of the factors influencing these levels of mechanical stress of the Essure® device implant will be assessed during tensile breakage and thermal breakage for its two parts (internal part and external part)
thermal resistance | During surgical intervention
  The thermal resistance of the Essure® device implant during coagulations/electrical sections will be assessed.
risk of degradation | During surgical intervention
  The risk of degradation depending on the temperature f the Essure® device implant used during coagulations/electrical sections will be assessed.
Concentrations of titanium constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of titanium constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of nickel constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of nickel constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of chromium constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of chromium constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of tin constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of tin constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of platinum constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of platinum constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of iridium constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of iridium constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of molybdenum constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of molybdenum constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of manganese constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of manganese constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of tungsten constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of tungsten constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of silver constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of silver constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
Concentrations of iron constituting the Essure® implant | up 12 months after surgical intervention
  Concentrations of iron constituting the Essure® implant in the peritoneal fluid, in the surgical piece, in the urine, in the blood, in the appendages (hair).
concentration of pro-inflammatory cytokines | Up 2 months after surgical intervention
  concentration of pro-inflammatory cytokines in the blood will be assessed
expression profile of miRNAs | Up 2 months after surgical intervention
  Expression profile of miRNAs in the peritoneal fluid will be assessed.
activated T lymphocyte profile | Up 2 months after surgical intervention
  activated T lymphocyte profile in blood will be assessed.
analysis of inflammatory pathway mRNAs | Up 2 months after surgical intervention
  analysis of inflammatory pathway mRNAs (nanostring® technology) in a pathology sample from the surgical specimen will be assessed.
Percentage of detection of Human Leukocyte Antigen | Up 2 months after surgical intervention
  Percentage of detection of Human Leukocyte Antigen (HLA)-DR53 (DRB4∗01) associated with nickel allergies in blood will be assessed.
Functional brain functions | up 6 months after Surgical intervention
  MRI-PET (Magnetic resonance imaging- Positron Emission Tomography) examination :
  * Mapping of brain inflammation: binding potential mapping of [11C]PK11195 characteristic of activated microglia
  * Brain anatomical imaging: clinical type anatomical MRI examination to assess the presence of cerebral anatomical abnormality
  * Brain mapping of functional connectivity at rest using Functional magnetic resonance imaging (fMRI)
  * Brain mapping of structural connectivity by diffusion MRI
  * Perfusion imaging : perfusion MRI examination without contrast product to assess the presence of cerebral perfusion abnormality
  * Magnetic susceptibility imaging: to detect possible hemorrhages

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU de Angers, Angers
  - Hôpital Femme Mère Enfant (Hospices Civils de Lyon), Bron
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Jeanne de Flandres, Lille
  - Hôpital de La Conception, Marseille
  - Institut Mère Enfant Alix de Champagne, CHU Reims, Reims
  - CHU de Rouen, Rouen
  - Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Paule de Viguier, CHU de Toulouse, Toulouse
  - Hôpital André Mignot, Centre Hospitalier de Versailles, Versailles